CLINICAL TRIAL: NCT03114826
Title: Study of the Impact of VEGF Polymorphism on the Development of Renal Carcinoma in Renal Transplant Patients
Acronym: VE-CART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0015
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Polymorphism; VEGF; Renal Carcinoma; Renal Transplantation
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal cell carcinoma in renal transplant patients
  Interventions: Genetic: To study the polymorphism of the gene encoding VEGF (rs699947) as a predictive marker

INTERVENTIONS:
Genetic: To study the polymorphism of the gene encoding VEGF (rs699947) as a predictive marker — Study the polymorphism of the gene encoding VEGF (rs699947) as a predictive marker of the occurrence of renal cell carcinoma in renal transplant patients.

SUMMARY:
Renal transplant patients have on average 3-5 times more risk of developing cancer than the general population. This rate can be increased up to 10 to 15 times in some type of cancer like kidney cancer. Among the identified risk factors, immunosuppressants and, in particular, calcineurin inhibitors (ciclosporin and tacrolimus) play a major role in increasing cancers apart from their depressant effects on the immune system.

Calcineurin inhibitors (CCN) are the basis of immunosuppressive therapy in renal transplantation. Several mechanisms have been implicated to explain their pro-oncogenic properties. One related to an increase in VEGF expression seems particularly interesting in the study of renal cell carcinoma in the transplanted patient. Indeed, the physiopathology of kidney cancer has clearly been associated with an increase in the production of VEGF. Furthermore, some polymorphisms of the gene encoding VEGF have already been associated with the survival of patients with renal carcinoma and the circulating level of VEGF in the general population. The search for an association between the polymorphisms of the VEGF gene and renal carcinoma in renal transplant patients could thus identify patients whose risk of renal cell carcinoma (cRCC) post-transplantation is increased. If the involvement of certain polymorphisms in the development of cRCC was confirmed in this population, their research before the introduction of the immunosuppressive treatment would make it possible to direct the choice of treatment towards molecules without pro-oncogenic property in the Patients such as mTOR protein inhibitors (sirolimus, everolimus). This research project is therefore in line with the desire to move towards a more "personalized" medicine that could be beneficial for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a first, second or third kidney transplant;
* Patients receiving a transplant from a living or deceased donor, irrespective of the immunological risk;
* Patients with health insurance coverage;
* Live or deceased patients for which genomic DNA is available.
* in cases : first diagnosis of native kidney cancer (histological type: papillary or clear cell)

Exclusion Criteria:

* Minor transplant patients;
* Patients transplanted before 1 January 2002;
* Patients monitored in the interregion, but transplanted to another center;
* Patients receiving a double graft (kidney plus other organ) or a bi-graft;
* Patients not accepting that their medical data be included in the register;
* Patients not accepting that their specimen be used for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Renal transplant patients for the period 1 January 2002 to 31 December 2011
Sampling Method: Non-Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2016-10-06 (Actual); Primary Completion 2019-10-05 (Estimated); Study Completion 2019-10-05 (Estimated)

PRIMARY OUTCOMES:
Taqman allelic discrimination analysis allows to define, for each polymorphism studied, three genotypes: wild homozygote (WT / WT), heterozygote (WT / M), mutated homozygote (M / M). The presence of renal carcinoma was previously confirmed on biopsy. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France